CLINICAL TRIAL: NCT01054651
Title: Open-label, Randomized Clinical Trial in Kenya to Determine the Effectiveness of Artesunate + Sulfamethoxypyrazine/Pyrimethamine Vs. Praziquantel in the Treatment of S. Mansoni in Children
Brief Title: A Randomised Trial of Artesunate-sulfamethoxypyrazine/Pyrimethamine Versus Praziquantel for the Treatment of S. Mansoni
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: Dafra Pharma (Industry)
Responsible Party: Dr Charles O. Obonyo, Kenya Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEMRI SSC 1582; DRD140 - S6.2008 (Other: DAFRA Pharma)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Schistosoma Mansoni
Keywords: Schistosoma mansoni; Praziquantel; Artesunate + Sulfamethoxypyrazine/pyrimethamine; Randomized open-label controlled clinical trial
MeSH Terms: conditions — Schistosomiasis | interventions — Pyrimethamine; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artesunate+Sulfamethoxypyrazine/pyrimethamine (Experimental)
  Interventions: Drug: Artesunate+Sulfamethoxypyrazine/pyrimethamine
- Praziquantel (Active Comparator)
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Artesunate+Sulfamethoxypyrazine/pyrimethamine
  Other Names: Co-arinate FDC
  Arms: Artesunate+Sulfamethoxypyrazine/pyrimethamine
Drug: Praziquantel
  Other Names: Biltricide
  Arms: Praziquantel

SUMMARY:
The purpose of this study is to determine the comparative efficacy of artesunate plus sulfamethoxypyrazine-pyrimethamine versus Praziquantel in the treatment of school children infected with S.mansoni in western Kenya.

DETAILED DESCRIPTION:
Schistosomiasis remains an important parasitic disease in the tropics, including Kenya. In the absence of a vaccine, the major control strategy is the reduction of morbidity by chemotherapy using Praziquantel. Evidence from laboratory studies and field trials continue to show that schistosome worms have developed reduced susceptibility to Praziquantel. These observations indicate the need for research to monitor the trends in efficacy of praziquantel and the need for research to develop novel antischistosomal drugs. Randomized controlled trials have also shown that Artemisinin derivatives (artesunate, artemether) have antischistosomal activity against S. mansoni, S. haematobium and S. japonicum. We propose to conduct an open-label, randomized trial to evaluate the comparative efficacy of artesunate plus sulfamethoxypyrazine-pyrimethamine versus Praziquantel in the treatment of 212 school children infected with S.mansoni in Rarieda district in western Kenya. To do this we will screen about 1000 school children by examination of stool for schistosome eggs. Eligible children will be randomized to receive either artesunate plus sulfamethoxypyrazine-pyrimethamine over 3 days or a single dose of Praziquantel. Four weeks after treatment, the participants will be assessed for cure and egg reduction.Our study may provide vital information regarding an alternative treatment for S. mansoni infection in children.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 15 years old
* Study participants appear healthy at enrollment, as assessed by the study clinician
* Suffering from S. mansoni infection, excreting eggs in stool
* Residing in Uyoma area, near Lake Victoria
* Able to receive oral treatment
* Parent/legal guardian gives informed written consent for the child to participate in the study
* Child assent to participate in study

Exclusion Criteria:

* Weighing more than 50 kg
* Pregnant or lactating at the time of the study
* Presence of infection with Plasmodium falciparum or other Plasmodium spp.
* Presence of severe illness, such as cerebral cysticercosis
* Signs of severe malnutrition (defined as children with weight/height ratio below 3 standard deviations or below 70% of the median of the WHO standardized reference values, or still with symmetrical oedema affecting both feet)
* Hypersensitivity to As, sulfonamides or PZQ.
* Use of another anti-malaria or anti-schistosomal drug during the study, or within 28 days before the administration of treatment.
* Previous participation in this study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Compare the cure rate between the two treatment arms | after 28 days

SECONDARY OUTCOMES:
Compare the proportion of children excreting schistosoma eggs between the two treatment arms | after 28 days
Compare the amount of eggs produced between the two arms | after 28 days
Compare the incidence of clinical and biological adverse events | after 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pauline N Mwinzi, PhD, Study Director — Kenya Medical Research Institute
Locations (1):
- KEMRI Centre for Global Health Research, Kisumu, Kenya

REFERENCES:
- [Derived] Obonyo CO, Muok EM, Mwinzi PN. Efficacy of artesunate with sulfalene plus pyrimethamine versus praziquantel for treatment of Schistosoma mansoni in Kenyan children: an open-label randomised controlled trial. Lancet Infect Dis. 2010 Sep;10(9):603-11. doi: 10.1016/S1473-3099(10)70161-4. Epub 2010 Aug 10. PMID 20705516